CLINICAL TRIAL: NCT00835250
Title: Prospective Randomized Clinical Trial Comparing Laparoscopic Cholecystectomy and Hybrid Natural Orifice Translumenal Endoscopic Surgery (NOTES)
Brief Title: Laparoscopic Cholecystectomy vs Hybrid Natural Orifice Translumenal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Son Llatzer (Other)
Responsible Party: Principal Investigator, Jose F. Noguera, Chief Department of Surgery, Hospital Son Llatzer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LLATZERNOTES-2
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Cholelithiasis
Keywords: Transvaginal cholecystectomy; NOTES; Minilaparoscopy; Endoscopic surgery; Cholecystectomy; Surgical translumenal endoscopic surgery; Transvaginal translumenal endoscopic surgery
MeSH Terms: conditions — Cholelithiasis | interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Laparoscopy (Active Comparator): Laparoscopic cholecystectomy
  Interventions: Procedure: Cholecystectomy
- Transumbilical (Experimental): Transumbilical endoscopic cholecystectomy
  Interventions: Procedure: Cholecystectomy
- Transvaginal (Experimental): Transvaginal endoscopic cholecystectomy
  Interventions: Procedure: Transvaginal hybrid NOTES cholecystectomy; Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Transvaginal hybrid NOTES cholecystectomy — Cholecystectomy performed by using a combination of working tools inserted through the entry port for the minilaparoscopy and the videogastroscope, inserted into peritoneal cavity by transvaginal approach. The gallbladder is removed transvaginally through the videogastroscope.
  Other Names: NOTES cholecystectomy; Transvaginal cholecystectomy
  Arms: Transvaginal
Procedure: Cholecystectomy — Extirpation of the gallbladder by a surgical procedure

SUMMARY:
The purpose of the study is to determine the feasibility of cholecystectomy made by a transvaginal approach with a NOTES procedure (natural orifice translumenal endoscopic surgery).

DETAILED DESCRIPTION:
Natural orifice transluminal endoscopic surgery (NOTES) makes it possible to perform intraperitoneal surgical procedures with a minimal number of access points in the abdominal wall. At the present time these procedures are hybrids. It is expected a better cosmetic result and lower incidence in parietal complications in front of laparoscopic cholecystectomy, but is necessary to investigate that these benefits should not be associated with complications of the new access to abdominal cavity.

Methods. Prospective randomized clinical series of 60 female patients with gallstones that underwent endoscopic surgery, 20 of them operated with conventional laparoscopic approach, 20 by transumbilical endoscopic approach and 20 of them by transvaginal endoscopic approach. Variables as surgical wound infection, urinary tract infection, evisceration, hernia, mortality and other complications will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 and under 65
* symptomatic cholelithiasis with an indication for performing laparoscopic surgery
* absence of any gynecological condition that could complicate the procedure (pelvic inflammatory disease or endometriosis)
* perforated hymen
* agreement on the patient's part not to use the vagina for two weeks after the surgery
* signed specific informed consent upon providing specific information about the new surgical approach.

Exclusion Criteria:

* age under 18 or over 65
* unperforated hymen
* presence of illness or condition with an increased risk of pelvic damage with transvaginal approach.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Parietal complications after surgery (infection and hernia) | One year

SECONDARY OUTCOMES:
Surgical pain. General complications. Patient's preferences. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Angel Cuadrado, MD PhD, Study Chair — Hospital Son Llàtzer
Locations (1):
- Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Result] Dolz C, Noguera JF, Martin A, Vilella A, Cuadrado A. [Transvaginal cholecystectomy (NOTES) combined with minilaparoscopy]. Rev Esp Enferm Dig. 2007 Dec;99(12):698-702. doi: 10.4321/s1130-01082007001200004. Spanish. PMID 18290693
- [Derived] Noguera JF, Cuadrado A, Dolz C, Olea JM, Garcia JC. Prospective randomized clinical trial comparing laparoscopic cholecystectomy and hybrid natural orifice transluminal endoscopic surgery (NOTES) (NCT00835250). Surg Endosc. 2012 Dec;26(12):3435-41. doi: 10.1007/s00464-012-2359-4. Epub 2012 May 31. PMID 22648123